CLINICAL TRIAL: NCT05830734
Title: Examining the Effect of Additional Injection of Freshly Collected Autologous Adipose Tissue to Bascom's Cleft Lift Surgery in the Treatment of Pilonidal Disease- a Randomized Controlled Trial
Brief Title: Injection of Freshly Collected Autologous Adipose Tissue Additional to Bascom's Cleft Lift Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Region Zealand (Other)
Responsible Party: Principal Investigator, Susanne Haas, MD PhD, assosciate professor, Randers Regional Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCTBCLAFI2022
Record Dates: First submitted 2023-01-06; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Pilonidal Disease

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will all receive BCL surgery and all have two small incisions in in the lumbar region with local anesthetic injection and compression bandages. Only the intervention group with have fatty cells harvested and injected in the surgical wound. The out comes assessor is blinded to which treatment has been given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCL surgery with fatty cell injection arm (Experimental): Patients will undergo BCL surgery and additionally have to small incisions made in the lumbar region from which 80 ml of fatty cells are harvested. After harvest local anesthetics are injected bilaterally and a compression bandage applied. The fatty cells are injected into the surgical wound before closure. All wounds are lateralized and close with a suction drain removed after 3 days
  Interventions: Other: injection of freshly collected adipose cells; Procedure: Bascoms Cleft lift procedure
- BCL surgery alone arm (Sham Comparator): Patients will undergo BCL surgery. Additionally two small incisions are made in the lumbar region, local anesthetics are injected bilaterally and a compression bandage applied. All wounds are lateralized and close with a suction drain removed after 3 days
  Interventions: Procedure: Bascoms Cleft lift procedure

INTERVENTIONS:
Other: injection of freshly collected adipose cells — A small incision is made bilaterally in the lumbar region. 2-300 ml of Ringer's acetate with 1 mg of added adrenaline is introduced with an infusion cannula fan-shaped into the subcutaneous adipose tissue on each side of the region.
  Adipose tissue is harvested for a total of approx. 80 ml. 20 ml Bupivacaine 5 mg/ml is distributed on each side of the lower back. The incisions are then closed with Steri-Strips and a compressive dressing is applied to reduce the risk of hematoma.
  The harvested adipose tissue then centrifuged in bulks of four at 1000 rpm. minute for 3 minutes. The liquid fraction is discarded. Using a three-way tap system, the adipose tissue is microfragmented between two 10 ml syringes by moving the contents back and forth at least 20 times. The adipose tissue is then distributed in 2 ml syringes for injection. A total of between 25 and 55 ml of usable adipose tissue will be harvested.
  Arms: BCL surgery with fatty cell injection arm
Procedure: Bascoms Cleft lift procedure — The procedure is carried out according to standardized principles previously decribed by Drs. John and Tom Bascom

SUMMARY:
In brief, the right management of complex or recurrent pilonidal disease (PD) is still controversial. In our institution we treat these conditions with Bascom's cleft lift surgery. Though this approach for most parts is beneficial, a large proportion of patients will suffer from prolonged post operative healing. We have published some positive results on treating non-healing postoperative wounds after cleft lift surgery with autologous fatty cell transplantation. The overall aim of the project is to investigate whether the addition of autologous fat cell transplantation in the surgical treatment of PD reduces the incidence of patients with prolonged postoperative healing. In a double-blinded randomized controlled clinical trial, we will investigate the effect of injections of freshly harvested autologous fatty cells in addition to Bascom's cleft lift operation versus Bascom's cleft lift operation alone.

DETAILED DESCRIPTION:
The overall aim of the project is to investigate whether the addition of autologous fatty cell transplantation in the surgical treatment of pilonidal disease (PD) reduces the incidence of patients with prolonged postoperative healing. In a double-blinded randomized controlled clinical trial, the investigators will investigate the effect of injections of freshly harvested autologous fatty cells in addition to Bascom's cleft lift operation versus Bascom's cleft lift operation alone.

The investigators hypothesize that addition of autologous fatty cell injection to Bascom's cleft lift operation for pilonidal disease will reduce the proportion of patients with poor postoperative healing compared to patients in the control group who are treated with Bascom's cleft lift operation alone.

The primary endpoint of this study is healing of the pilonidal lesion (max 1 defect ≤5mm, no undermining) after 4 weeks and 12 weeks.

Further, symptom development, postoperative pain, complication rate, time to healing and recurrence rates are also explored.

BRIEF LITERATURE REVIEW:

Pilonidal disease (PD) is a widespread disorder that occurs in the crena ani. A paradigm shift in our perception of the pathology causing this disorder has been coming for several decades and the treatment is slowly conforming to this.

The estimated incidence is 26-48 per 100,000, although globally there is great geographical variation (1). Men present with treatment-requiring pilonidal disease more than twice as often as women, and population studies of young students have found up to a 10:1 male/female ratio, including asymptomatic pilonidal cysts(2). In the investigators own material, the proportion of women are 17% of patients with complicated pilonidal disease (62/363). The disorder most often affects younger patients with an average age at first manifestation of 21 years for men and 19 for women (1).

Acute manifestations are infected cysts and results in the formation of pilonidal abscesses. The treatment of these is uncontroversial and is based on lateral incision and drainage with secondary open healing.

Chronic pilonidal disease manifests itself in the formation of more or less widespread subcutaneous branching systems containing hair which is "sucked" into the system by negative pressure that occurs when changing position, especially from sitting to standing. The condition is characterized by pain and foul-smelling secretions and bleeding.

The treatment of the chronic manifestations, as opposed to the acute abscesses, has been controversial and over the last 1-2 decades has gradually moved more towards lateralization techniques, the gap between the buttocks is (partially) levelled surgically and the suture line is placed outside the midline of the crena ani (3,4).

Bascom's cleft lift operation is one of several lateralization techniques that have shown promising results over the past decades (5-10). Nevertheless, in the hands of the investogators poor or delayed healing is found in up to a third of these otherwise young and healthy patients, which seems to be in line with the international literature (11). Many patients thus experience long outpatient courses postoperatively with several additional treatments such as regular surgical wound revision, treatment with various forms of negative pressure bandaging, steroid cream regimens or silvernitrate dressings.

Platelet-rich plasma therapy (BPT) is used with good effect as an addition to the surgical treatment of pilonidal disease, as BPT promotes angiogenesis, cell regeneration and thus promotes healing. A review finds a reduction in healing time of 36% in BPT-treated patients compared to the control group(12,13). Moreover, treatments with allogeneic adipose-derived stem cells are used in other healing-challenged areas, such as mb. Crohn's fistulas and burns (14-16). However, both treatments are both time-consuming and expensive, and the investigators believe that autologous fat cell transplantation is a faster and more affordable alternative, which a study in Mb. Crohn's patients with complicated peri-anal fistulas also support: Here, in a series of 21 patients healing was found in 57% (clinical and MR-verified) - a very satisfactory result in this context (17). The cell composition in the stromal vascular fraction (SVF) of the harvested adipose tissue has been found to contain 10%-50% live stromal (mesenchymal) stem cells and 7%-30% endothelial cells (mature and stem cells) depending on where the fat is harvested and which method is used (18-20). This cell composition supports the healing potential in the treatment with autologous fatty cell transplantation.

In the department of the investigators, a series of operations with autologous fatty cell injections for non-healing pilonidal wounds has been carried out with good results. Thus, in these highly selected patients, the investigators have a healing rate of 83% (69-96%) over a median time of 159 days. Two patients had recurrence (6.7%) (21).

The method is minimally invasive and is combined in this study with Bascom's cleft lift (BCL) operation. The results seem promising with minimal risks and it could be an important supplement to the basic treatment of these patients.

3) METHOD

STUDYDESIGN:

The study will be conducted as a double-blinded randomized controlled clinical trial that will compare healing after BLC surgery with injections of freshly harvested autologous adipose tissue versus BLC surgery alone. The trial is being conducted as a multicenter study, where patients are included at two centers in Denmark. The two centers are located at Randers Regional Hospital and Slagelse Hospital.

SURGICAL PROCEDURE:

Included patients will undergo BLC surgery according to standardized principles. Prior to surgery, the randomization is carried out using allocation tables in REDCap, where an equal distribution of patients in the intervention group and the control group is also ensured in each center.

Intervention group: Patients in the intervention group will undergo liposuction to harvest autologous fatty cells. The patient is placed in prone position. For the liposuction, a small incision is made bilaterally in the flanks. 2-300 ml of Ringer's acetate with 1 mg of added adrenaline is introduced with an infusion cannula fan-shaped into the subcutaneous adipose tissue on each side of the lumbar region.

Adipose tissue is harvested with an equal distribution on each side of the region for a total of approx. 80 ml. 20 ml Bupivacaine 5 mg/ml is distributed on each side of the lower back after harvesting the fatty cells. The incisions are then closed with Steri-Strips and a compressive dressing is applied to reduce the risk of hematoma.

The adipose tissue is then prepared: The harvested adipose tissue is distributed equally in 10 ml syringes and centrifuged in bulks of four at 1000 rpm. minute for 3 minutes. The liquid fraction is discarded. Using a three-way tap system, the adipose tissue is homogenized/microfragmented between two 10 ml syringes by moving the contents back and forth at least 20 times. The adipose tissue is then distributed in 2 ml syringes for injection. A total of between 25 and 55 ml of usable adipose tissue will be harvested.

Bascom cleft lift operation is performed as described in appendix 7. Before the cleft lift incision is sutured, the fatty tissue will be systematically injected with a sharp 1.2 mm needle and cover all the wound surfaces with 0.2-0.5 ml at a time. The procedure was published as a video vignette in 2019(22). Results from the first seven patients (2020) and the first 30 patients (2022) have been published (21,23).

Patients in the control group: Control patients are given a sham, where a small incision is also made bilaterally in the lumbar region and 20 ml Bupivacaine 5 mg/ml is distributed on each side of the lower back. The incisions are then closed with Steri-Strips and compressive dressings are applied in the same way as the intervention group.

COOPERATION PARTNERS:

Surgeries will be performed by specialists in abdominal surgery with a sub-specialty within this type of surgery in two centres: Surgical Department at Randers Regionshospital and Slagelse Hospital. I. Faurschou at Randers Regionshospital, Region Midt, has the overall responsibility for the project with Supervisor Susanne Haas as the legally responsible person. The local manager at Slagelse Hospital is P. Maine. Those responsible at each site are responsible for inclusion and informing the patients, guided and supported by I. Faurschou.

POST-OPERATIV FOLLOW-UP:

The patients will have follow ups at 4 and 12 weeks after the operation, where the healing will be clinically assessed based on endpoints by project manager I. Faurschou, blinded to the randomisation. The control takes place by telephone consultation together with answering the symptom questionnaire and pain diary sent out automatically from REDCap® as well as weekly photo documentation of healing through Pleje.net® (Dansk Telemedicin A/S), with the option of immediate physical consultation within a week in case of lack of healing. Photos will be taken using the Pleje.net app weekly in relation to hair removal by a nurse/person who handles hair removal. Patients are given a guide to Pleje.net. On Pleje.net, a user group has been set up for each site, so only project managers can see all the patients.

If there is no healing after 12 weeks, the patient will be offered further treatment in line with our normal treatment practice.

4) STATISTICAL CONSIDERATIONS:

Sample size: In a recent study, the investigators found somewhat surprisingly that only 12% of PS patients operated with BCL surgery were fully healed after 14 days (≤ 1 defect, ≤ 5 mm, no undermining). After 12 weeks, this proportion was 72%. The investigaros expect 50% of patients to have healed after 4 weeks.

Using fatty cells in non-healing PS wounds, the investigators have a healing rate of 83% (69-96%) over a median time of 159 days. In combination with fatty cells, it is expected that 75% of patients have healed by 4 weeks. With a significance level of 5% (α) and a power of 80% (β), 66 patients will be included in each group (Fleiss with continuity correction). Assuming a dropout of 4 patients in each group, a total of 140 patients will be included.

Interim analysis: Interim analysis: Halfway through the inclusion, an interim analysis will be carried out. A Data Monitoring Committee (DMC) is set up, which will make a recommendation to the project managers on whether the study should continue as planned, be interrupted due to unintended side effects as a result of AFT, interrupted because the effect of AFT has been unequivocally established; or is interrupted because it will not be possible to see a difference if the study is continued.

5) PATIENTS: The patients are referred to the investigators outpatient clinic and informed about the project if BCL surgery is needed (recurrent or complex disease). After reflection time, patients are included on the day of surgery, where they are randomised. After the operation, they will be followed in the outpatient 4 weeks and 12 weeks postoperatively. If there is no healing after 12 weeks, the patient will be offered further treatment in line with our normal treatment practice.

ELIGIBILITY:
Inclusion Criteria:

Advanced pilonidal disease with indication for surgery with Bascom's cleft lift surgery due to either

1. Primary extensive manifestation where minimally invasive surgery is not possible
2. Lack of healing after previous surgery (> 2 months)
3. Recurrence after previous elective surgery

   * Informed and written consent, as well as consent for follow-up.
   * Danish speaking/reading and thus able to understand Danish patient information, questionnaires and the pleje.net system.

Exclusion Criteria:

* Acute infection in pilonidal disease
* Pregnancy
* BMI <20 and >35
* Smokers (stop smoking at least 6 weeks before and after the operation)
* Insulin-dependent diabetes
* Age <15 years
* Bilateral extension not suitable for BCL surgery

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
healing | 4 weeks
  Healing of the pilonidal lesion (max 1 defect ≤5mm, no undermining)
healing | 12 weeks
  Healing of the pilonidal lesion (max 1 defect ≤5mm, no undermining)

SECONDARY OUTCOMES:
Symptom development | pre-operatively, at 4 weeks, 12 weeks and 12 months
  Symptom questionnaire completed .
postoperative pain | first 14 postoperative days
  pain diary. Daily pain measurement on a VAS score (0= no pain, 10= worst imaginable pain)
complications | 12 weeks
  any early or late complications that may arise
Time to healing | upto 12 months
  the patients will be followed weekly with photos in pleje.net until healing has occured
recurrence | 12 months
  recurrent disease after complete healing is registered by questionnaire
recurrence | 36 months
  recurrent disease after complete healing is registered by questionnaire
recurrence | 60 months
  recurrent disease after complete healing is registered by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: susanne Haas, MD PHD, Study Chair — University of Aarhus
Locations (1):
- Regions Hospitalet Randers, Randers, Jylland, Denmark

IPD SHARING:
Plan to Share IPD: No
we will share individual participant data if necessary in the reviewing process

REFERENCES:
- [Background] Sondenaa K, Andersen E, Nesvik I, Soreide JA. Patient characteristics and symptoms in chronic pilonidal sinus disease. Int J Colorectal Dis. 1995;10(1):39-42. doi: 10.1007/BF00337585. PMID 7745322
- [Background] Luedi MM, Schober P, Stauffer VK, Diekmann M, Doll D. Global Gender Differences in Pilonidal Sinus Disease: A Random-Effects Meta-Analysis. World J Surg. 2020 Nov;44(11):3702-3709. doi: 10.1007/s00268-020-05702-z. Epub 2020 Jul 17. PMID 32681319
- [Background] Enriquez-Navascues JM, Emparanza JI, Alkorta M, Placer C. Meta-analysis of randomized controlled trials comparing different techniques with primary closure for chronic pilonidal sinus. Tech Coloproctol. 2014 Oct;18(10):863-72. doi: 10.1007/s10151-014-1149-5. Epub 2014 Apr 30. PMID 24845110
- [Background] McCallum IJ, King PM, Bruce J. Healing by primary closure versus open healing after surgery for pilonidal sinus: systematic review and meta-analysis. BMJ. 2008 Apr 19;336(7649):868-71. doi: 10.1136/bmj.39517.808160.BE. Epub 2008 Apr 7. PMID 18390914
- [Background] Bascom J, Bascom T. Failed pilonidal surgery: new paradigm and new operation leading to cures. Arch Surg. 2002 Oct;137(10):1146-50; discussion 1151. doi: 10.1001/archsurg.137.10.1146. PMID 12361421
- [Background] Bascom J, Bascom T. Utility of the cleft lift procedure in refractory pilonidal disease. Am J Surg. 2007 May;193(5):606-9; discussion 609. doi: 10.1016/j.amjsurg.2007.01.008. PMID 17434365
- [Background] Guner A, Boz A, Ozkan OF, Ileli O, Kece C, Reis E. Limberg flap versus Bascom cleft lift techniques for sacrococcygeal pilonidal sinus: prospective, randomized trial. World J Surg. 2013 Sep;37(9):2074-80. doi: 10.1007/s00268-013-2111-9. PMID 23732258
- [Background] Iesalnieks I, Deimel S, Schlitt HJ. Karydakis flap for recurrent pilonidal disease. World J Surg. 2013 May;37(5):1115-20. doi: 10.1007/s00268-013-1950-8. PMID 23435676
- [Background] Nordon IM, Senapati A, Cripps NP. A prospective randomized controlled trial of simple Bascom's technique versus Bascom's cleft closure for the treatment of chronic pilonidal disease. Am J Surg. 2009 Feb;197(2):189-92. doi: 10.1016/j.amjsurg.2008.01.020. Epub 2008 Jul 17. PMID 18639221
- [Background] Theodoropoulos GE, Vlahos K, Lazaris AC, Tahteris E, Panoussopoulos D. Modified Bascom's asymmetric midgluteal cleft closure technique for recurrent pilonidal disease: early experience in a military hospital. Dis Colon Rectum. 2003 Sep;46(9):1286-91. doi: 10.1007/s10350-004-6729-4. PMID 12972977
- [Background] Iesalnieks I, Ommer A. The Management of Pilonidal Sinus. Dtsch Arztebl Int. 2019 Jan 7;116(1-2):12-21. doi: 10.3238/arztebl.2019.0012. PMID 30782310
- [Background] Mostafaei S, Norooznezhad F, Mohammadi S, Norooznezhad AH. Effectiveness of platelet-rich plasma therapy in wound healing of pilonidal sinus surgery: A comprehensive systematic review and meta-analysis. Wound Repair Regen. 2017 Nov;25(6):1002-1007. doi: 10.1111/wrr.12597. Epub 2018 Feb 7. PMID 29215166
- [Background] Mohamadi S, Norooznezhad AH, Mostafaei S, Nikbakht M, Nassiri S, Safar H, Moghaddam KA, Ghavamzadeh A, Kazemnejad A. A randomized controlled trial of effectiveness of platelet-rich plasma gel and regular dressing on wound healing time in pilonidal sinus surgery: Role of different affecting factors. Biomed J. 2019 Dec;42(6):403-410. doi: 10.1016/j.bj.2019.05.002. Epub 2019 Dec 10. PMID 31948604
- [Background] Cabalzar-Wondberg D, Turina M, Biedermann L, Rogler G, Schreiner P. Allogeneic expanded adipose-derived mesenchymal stem cell therapy for perianal fistulas in Crohn's disease: A case series. Colorectal Dis. 2021 Jun;23(6):1444-1450. doi: 10.1111/codi.15587. Epub 2021 Mar 5. PMID 33595166
- [Background] Garcia-Arranz M, Herreros MD, Gonzalez-Gomez C, de la Quintana P, Guadalajara H, Georgiev-Hristov T, Trebol J, Garcia-Olmo D. Treatment of Crohn's-Related Rectovaginal Fistula With Allogeneic Expanded-Adipose Derived Stem Cells: A Phase I-IIa Clinical Trial. Stem Cells Transl Med. 2016 Nov;5(11):1441-1446. doi: 10.5966/sctm.2015-0356. Epub 2016 Jul 13. PMID 27412883
- [Background] Chang YW, Wu YC, Huang SH, Wang HD, Kuo YR, Lee SS. Autologous and not allogeneic adipose-derived stem cells improve acute burn wound healing. PLoS One. 2018 May 22;13(5):e0197744. doi: 10.1371/journal.pone.0197744. eCollection 2018. PMID 29787581
- [Background] Dige A, Hougaard HT, Agnholt J, Pedersen BG, Tencerova M, Kassem M, Krogh K, Lundby L. Efficacy of Injection of Freshly Collected Autologous Adipose Tissue Into Perianal Fistulas in Patients With Crohn's Disease. Gastroenterology. 2019 Jun;156(8):2208-2216.e1. doi: 10.1053/j.gastro.2019.02.005. Epub 2019 Feb 14. PMID 30772343
- [Background] Astori G, Vignati F, Bardelli S, Tubio M, Gola M, Albertini V, Bambi F, Scali G, Castelli D, Rasini V, Soldati G, Moccetti T. "In vitro" and multicolor phenotypic characterization of cell subpopulations identified in fresh human adipose tissue stromal vascular fraction and in the derived mesenchymal stem cells. J Transl Med. 2007 Oct 31;5:55. doi: 10.1186/1479-5876-5-55. PMID 17974012
- [Background] Zimmerlin L, Donnenberg VS, Pfeifer ME, Meyer EM, Peault B, Rubin JP, Donnenberg AD. Stromal vascular progenitors in adult human adipose tissue. Cytometry A. 2010 Jan;77(1):22-30. doi: 10.1002/cyto.a.20813. PMID 19852056
- [Background] Yoshimura K, Shigeura T, Matsumoto D, Sato T, Takaki Y, Aiba-Kojima E, Sato K, Inoue K, Nagase T, Koshima I, Gonda K. Characterization of freshly isolated and cultured cells derived from the fatty and fluid portions of liposuction aspirates. J Cell Physiol. 2006 Jul;208(1):64-76. doi: 10.1002/jcp.20636. PMID 16557516
- [Background] Sophie VG, Marlene SJ, Helene HT, Lilli L, Allan PG, Susanne H. Injection of freshly collected autologous adipose tissue in complicated pilonidal disease: a prospective pilot study. Tech Coloproctol. 2022 Nov;26(11):883-891. doi: 10.1007/s10151-022-02683-0. Epub 2022 Aug 13. PMID 35963978
- [Background] Elfeki H, Sorensen MJ, Pedersen AG, Lundby L, Haas S. Injection of freshly collected autologous adipose tissue for treatment of a non-healing sacrococcygeal pilonidal disease patient - a video vignette. Colorectal Dis. 2019 Nov;21(11):1341. doi: 10.1111/codi.14806. Epub 2019 Aug 23. No abstract available. PMID 31389100
- [Background] Haas S, Sorensen MJ, Lundby L, Pedersen AG. Injection of freshly collected autologous adipose tissue into non-healing wounds after closed incision pilonidal surgery. Tech Coloproctol. 2020 Dec;24(12):1301-1306. doi: 10.1007/s10151-020-02276-9. Epub 2020 Jul 9. PMID 32648140